CLINICAL TRIAL: NCT03941756
Title: Prophylactic Lymphovenous Bypass Procedure Following Axillary Lymphadenectomy: A Prospective Observational Study
Brief Title: Lymphovenous Bypass Procedure Before Underarm Lymph Node Surgery in Preventing Lymphedema in Patients With Inflammatory or Locally Advanced Non-inflammatory Breast Cancer or Melanoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0127; NCI-2019-02320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0127 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Breast Inflammatory Carcinoma; Locally Advanced Breast Carcinoma; Melanoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Melanoma | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (LVB) (Experimental): Patients receive indocyanine green IV and undergo lymphangiography, then undergo LVB at the time of ALND.
  Interventions: Drug: Indocyanine Green; Procedure: Lymphangiography; Procedure: Lymphovenous Bypass
- Group II (no intervention) (No Intervention): Patients do not receive indocyanine green, undergo lymphangiography, nor undergo LVB at the time of ALND.

INTERVENTIONS:
Drug: Indocyanine Green — Given IV
  Other Names: ICG
  Arms: Group I (LVB)
Procedure: Lymphangiography — Undergo lymphangiography
  Other Names: Lymphography
  Arms: Group I (LVB)
Procedure: Lymphovenous Bypass — Undergo LVB
  Other Names: Lymphovenous Anastomosis
  Arms: Group I (LVB)

SUMMARY:
This pilot trial studies whether a procedure called lymphovenous bypass would prevent lymphedema (arm swelling) in patients with inflammatory breast cancer or non-inflammatory breast cancer that has spread to nearby tissues or lymph nodes or melanoma. The lymphovenous bypass procedure creates a path for lymphatic fluid to flow away from the arms. It is usually done after a diagnosis of lymphedema. In this study, giving lymphovenous bypass before underarm lymph node surgery may help prevent lymphedema from forming.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the protective benefit to performing standard of care lymphovenous bypass (LVB) surgery at the time of standard of care axillary lymph node dissection (ALND) for patients that are high risk for developing breast-cancer related lymphedema (LE) of the upper extremity.

SECONDARY OBJECTIVES:

I. Compare the medical outcomes for patients that received the LVB surgery with those receiving standard surgery in whom the intervention could not be performed.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive indocyanine green intravenously (IV) and undergo lymphangiography, then undergo LVB at the time of ALND.

GROUP II: Patients do not receive indocyanine green, undergo lymphangiography, nor undergo LVB at the time of ALND.

After completion of study, patients are followed up at 2 weeks, and then at 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years of age.
* Patients willing to participate.
* Patients able to complete informed consent.
* Patients will be eligible for inclusion if they fall into one for two groups:

  * Patients with inflammatory breast cancer, and those with locally advanced non-inflammatory breast cancer that are undergoing ALND and are anticipated to receive radiation therapy
  * Or: Patients with a diagnosis of melanoma (including unknown primary) that will undergo ALND will also be eligible for inclusion in the study as a comparator group.

Exclusion Criteria:

* Patients taking anticoagulants within 7 days prior to surgery.
* Patients that are known to be pregnant at the time of surgery.
* Patients are available for follow-up less than 18 months or do not undergo measurements within the scheduled period.
* Patients with body mass index (BMI) greater than 50.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Volumetric diagnosis of lymphedema | 18 months
  If the limb volume change, meets the criteria for a diagnosis of lymphedema at any time (5 percent, change), then the patient receives a diagnosis of lymphedema.
Incidence of lymphedema | 18 months
  Will compare the incidence of lymphedema after mastectomy and axillary lymph node dissection surgery between two surgical techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schaverien, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States